CLINICAL TRIAL: NCT04272281
Title: Utilisation d'un Outil de décision médicale partagée Dans la Prise en Charge Des Cystites Aigues Sans Risque de Complication en médecine générale : Comparaison de la Consommation d'Antibiotique Entre Deux Groupes randomisés en Cluster.
Brief Title: Use of a Share Decision Making Tool in the Care of Acute Cystitis Without Risk of Complication in Primary Care
Acronym: ARIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/48
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Cystitis
Keywords: primary health care; share decision making; antibiotics; daily activities
MeSH Terms: conditions — Cystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Share making tool decision (Experimental): Patient recruited from general practitioner in this group will use a share making tool decision to adapt antibiotherapy
  Interventions: Procedure: medical shared decision
- Standard recommandation (Active Comparator): Patients recruited from general practitioner will receive the standard medical care
  Interventions: Procedure: Standard medical care

INTERVENTIONS:
Procedure: medical shared decision — The experimental group will use the share decision making tool during consultation to adapt antibiotherapy
  Arms: Share making tool decision
Procedure: Standard medical care — control group will act as usual in their practice.
  Arms: Standard recommandation

SUMMARY:
the aim of this trial is to demonstrate that when caring women with symptoms of acute cystitis without any risk of complication, general practitioner may use share decision making tool to help patients better understand the stakes of taking antibiotics.

DETAILED DESCRIPTION:
Each year, more than 2.000.000 patients visit their general practitioners for a acute cystitis. The scientific literature shows that acute cystitis without risk of complication cause complications, such as pyelonephritis, in a very rare cases. However, French guidelines systematically request an antibiotic therapy as soon as the diagnostic is confirmed with the only goal to lowering symptomatology.

Recent studies show that some informed women would like not to take antibiotics and pain-killers could be as effective as antibiotics. Canadian studies assessing share decision making tools in patients with acute respiratory infection have shown that matching antibiotic treatment with the patient values lower such prescription without any impact on clinical outcomes .

Investigators aim to assess a similar strategy in patients with acute cystitis. This study will compare a group following French guidelines versus one using a share decision making tool to determine if, after being informed of the benefice and risk of this treatment, patient still want an antibiotic. Targeting instead of systematic prescription will reduce antibiotic consumption.

After diagnostic of acute cystitis to a woman between 18 and 65 years, investigators check if they filing all study criteria and ask for authorization to add them to the study. Then they'll act following their group instruction, and get information (antibiotic prescription or not, score to the Activity Impairment Assessment (AIA) scale, Score to satisfaction scale). Then patients will be followed by phone contact on day 5, day 14 and day 90 after inclusion to get information on antibiotic use, AIA and satisfaction scores and clinical outcomes, such urinary infection. Data on antibiotics delivery by pharmacy will be obtained through National assurance database.

ELIGIBILITY:
Inclusion Criteria:

* woman
* between 18 and 65 years
* symptom of acute cystitis without risk of complication
* affiliated to the French public welfare system
* with signed consent

Exclusion Criteria:

* anomaly of the urinary canal
* pregnancy
* more than 3 cystitis during the last year
* cancer, immunosuppression
* hemopathy, fever
* back-pain
* severe renal failure
* refuse to give consent and previously participate to the study
* under guardianship

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 169 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Use of antibiotic for acute cystitis without risk of complication | Day 14 after inclusion (day 0)

SECONDARY OUTCOMES:
Score at the "Activity Impairment Assessment" scale | Day 0, Day 5 and Day14
  Scale from 0 (never) to 4 (always) on several items about usuals activities limitations.
Score at the satisfaction scale | Day 0, Day 5, Day14 and Day 90
  Scale from 0 (not satisfied) to 10 (very satisfied) on satisfation about medical care.
Recurrence of the infection | Between Day 15 and Day 90
  Infection reccurence will be assessed with the number of dispensation of antibiotics between day 15 and day 90.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No